CLINICAL TRIAL: NCT02680106
Title: EVALUATION OF THE SPINNER™ DEVICE FOR THE APPLICATION OF WOUND DRESSING: TREATMENT OF SPLIT SKIN-GRAFT DONOR SITES. A Prospective, Safety and Efficacy, Open Labeled, Two Arms, Randomized, Multi Center, Controlled Study
Brief Title: Evaluation of the SPINNER Device for the Application of Wound Dressing: Treatment of Split Skin Graft Donor Sites
Acronym: SPINNER01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanomedic Technologies Ltd. (Industry)
Responsible Party: Sponsor
Organization: Nicast Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP0007
Record Dates: First submitted 2016-02-01; First posted 2016-02-11 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2019-03

CONDITIONS: Wound of Skin
Keywords: Nanofibers; Dressing; Donor site; Polycaprolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPINNER (Experimental): All patients in this arm will be treated with the SPINNER .
  Interventions: Device: SPINNER
- JELONET or IBU-Biatain (Active Comparator): All patients in this arm will be treated with JELONET/IBU Biatain dressing, regarded as the standard of current care for split-skin donor-site wounds.
  Interventions: Device: JELONET / IBU Biatain

INTERVENTIONS:
Device: SPINNER — The SPINNER device is aimed at the DSW from a distance of 20 cm and activated for 1 minute. A nano-fibrous matrix is thus created.
  Arms: SPINNER
Device: JELONET / IBU Biatain — The patient's DSW will be dressed by JELONET/IBU Biatain
  Arms: JELONET or IBU-Biatain

SUMMARY:
Evaluation of safety and performance of the SPINNER device and wound dressing in the treatment of donor-site wounds (DSW)

DETAILED DESCRIPTION:
The SPINNER is a hand held, portable electro-spinning device that produces personalized in-situ nanofiber dressings for the treatment of external burns and wounds.

The dressing has non-adherence, high absorbance, bacterial protection, easy and pain-free peel characteristics and shows excellent conformability and optimal coverage of the wound.

The objective of this study is to evaluate the safety and performance of the SPINNER device and wound dressing in the treatment of donor-site wounds (DSW) at size of 10-200 cm2.

The study will include five sites in Israel:

Sheba Medical Center, Tel Hashomer RambamMedical Center, Haifa Kaplan Medical Center, Rehovot Souraski Medical Center, Tel Aviv Beilinson Medical Center, Petach Tikva

Study primary endpoints:

1. Dermal Safety
2. Wound healing and time to complete re-epithelialization at 1, 3, 5, 7, 14 and 21 days post operation

Study secondary endpoints:

1. Ease of use
2. Pain assessment at 1, 3, 5, 7, 14 and 21 days post operation
3. Infection assessment from 3 days post operation up to 21 days
4. Device related adverse events of the SPINNER device and wound dressing

Extended exploratory follow up:

Assessment of itching and scarring from wound closure time and up to 12 months follow up

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥ 18 years old at enrolment. Both genders.
* Patients with donor site wound, size of 10-200 cm2, located in the thigh after partial thickness skin-graft
* The patient is able and willing to comply with study procedures and give written informed consent prior to enrollment in the study

Exclusion Criteria:

* Any known or suspected systemic infection
* Any known sensitivity to components/products used in this study
* Use of penicillamine, corticosteroid or immunosuppressive medication within two months prior to enrollment, or current use of nonsteroidal anti- inflammatory agents which cannot be discontinued, or who is likely to be prescribed these medications or any other medications known to adversely affect wound healing during study participation
* Major uncontrolled systemic disorders such as hepatic, renal, neurologic, or endocrinologic disorders.
* Patients undergoing repeat skin graft harvesting at the same donor site
* Patients with burns of more than 15% TBSA
* Requires immersion hydrotherapy at any time during study participation
* Bleeding disorders
* Skin disorders such as psoriasis, pemphigus, Toxic Epidermal Necrolysis (TEN), Stevens-Johnson Syndrome (SJS), pyoderma gangrenosum and other exfoliative disorders
* Terminal patients
* Soldiers
* Prisoners
* Female patients who are pregnant or nursing, or of childbearing potential and are not using adequate contraception
* Participation in another clinical trial within 30 days prior to the Screening Visit or during this study.
* Psychiatric patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in dermal safety (Draize) score | 1-21 days
  Change in Draize score from procedure day to day 21
Change in wound healing | 1-21 days
  Change in wound healing in cm2 from procedure day to day 21

SECONDARY OUTCOMES:
Ease of use | 21 days
  Ease of use will be assessed (questionnaire) by the users whenever the SPINNER is used.
Assessment of pain | 21 days
  Assessment of pain (VAS scale 0-10) at 1, 3, 5, 7, 14 and 21 days post operation.
Assessment of infection | 21 days
  Assessment of infection (questionnaire) from 3 days post operation up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Moti Harats, MD, Principal Investigator — Sheba Medical Center
Locations (5):
- Israel (5):
  - Rambam Medical Center, Haifa
  - Beilinson Medical Center, Petah Tikva
  - Burn Unit, Sheba Medical Center, Ramat Gan
  - Kaplan Hospital, Rehovot
  - Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No